CLINICAL TRIAL: NCT04199611
Title: Validating Clinical Efficacy for Integrated Psychological Intervention for Obesity: Physical Therapy and Psychotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Global 365MC Hospital (Unknown)
Responsible Party: Principal Investigator, Hyung Jin Choi, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-1811-124-990
Record Dates: First submitted 2019-12-10; First posted 2019-12-16 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Mental Health Issue; Body Image
Keywords: Body Image Satisfaction; Liposuction; Psychological Therapy
MeSH Terms: interventions — Lipectomy; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Integrated Therapy Group (Experimental): Both liposuction and psychological therapy are delivered to the participants in this group.
  Interventions: Procedure: Liposuction; Behavioral: Cognitive Behavioral Therapy
- Liposuction Group (Active Comparator): This group experiences only liposuction and do self-help care after the liposuction.
  Interventions: Procedure: Liposuction
- Psychological Therapy Group (Active Comparator): This group experiences only cognitive behavioral therapy (CBT; psychological therapy) during the intervention period.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Self-help Group (No Intervention): This group do not receive any interventions and do self-help care.

INTERVENTIONS:
Procedure: Liposuction — This is a type of fat removal procedure used in plastic surgery.
  Arms: Integrated Therapy Group; Liposuction Group
Behavioral: Cognitive Behavioral Therapy — This is a psycho-social intervention that aims to improve mental health.
  Other Names: CBT
  Arms: Integrated Therapy Group; Psychological Therapy Group

SUMMARY:
This study is to develop an integrated therapy (physical therapy and psychotherapy) to treat cognitive distortion for body image. Then, validate its efficacy to make an improvement in both physical and mental health.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25~30
* The score over 68 in SIMS (The situational motivation scale)

Exclusion Criteria:

* Diagnosed in any chronic disease
* Trouble using smartphone
* Pregnant or planning to be pregnant
* Unable to be in the fMRI
* Limited to be involved in physical activities over 30 minutes
* already had an experience in liposuction

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
BSQ-8C | 4 weeks, 8-item, scale 1 through 6
  Body Shape Questionnaire

SECONDARY OUTCOMES:
fMRI | 24 hours
  Brain response to the task-based fMRI
Computerized cognitive behavioral task | 24 hours
  dot-probe task and implicit association task
KoQoL | 24 hours, 13-item, scale 1 through 4
  Korean version of Obesity-related Quality of Life
DEBQ | 24 hours, 33-item, scale 1 through 5
  Dutch Eating Behavioral Questionnaire
K-BDI | 24 hours, 21-item, scale 1 through 4
  Korean Beck Depression Inventory
RSES | 24 hours, 10-item, scale 1 through 4
  Rosenberg Self Esteem Scale
TAI | 24 hours, 20-item, scale 1 through 4
  Trait Anxiety Inventory
PANAS | 24 hours, 20-item, scale 1 through 5
  Positive and Negative Affect Schedule
SCL-90-R | 24 hours, 90-item, scale 1 through 5
  The Symptom Checklist-90-R
EAT-26 | 24 hours, 26-item, scale 1 through 6
  The Eating Attitudes Test 26
K-AAQ-II | 24 hours, 10-item, scale 1 through 7
  Korean version of The Acceptance and Action Questionnaire - II
Cognitive bias on the body image | 24 hours, one-item, scale 1 through 4
  What do you think about your body image based on the BMI criteria?
BMI in kg/m^2 | 24 hours
  body weight and height
Body fat percent | 24 hours
  the total mass of fat divided by total body mass, multiplied by 100
Leg circumference | 24 hours
  locating the biggest part of your upper leg
Waist circumference | 24 hours
  a measurement taken around the abdomen at the level of the umbilicus.
Glucose | 24 hours
  blood sample
ALT | 24 hours
  Alanine transaminase
AST | 24 hours
  Aspartate transaminase
GGT | 24 hours
  Gamma-glutamyltransferase
Total Cholesterol | 24 hours
  blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Meelim Kim, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Clinical Study Report (CSR)